CLINICAL TRIAL: NCT03678571
Title: Latrunculin A for Oocyte Vitrification
Brief Title: Oocyte Vitrification Aided With Latrunculin A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banoon IVF Center (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSina-Oocyte-LA
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latrunculin A supplemented vitrification medium (Experimental)
  Interventions: Other: Latrunculin A supplemented vitrification medium
- Vitrification medium with no supplementation (No Intervention)

INTERVENTIONS:
Other: Latrunculin A supplemented vitrification medium — Vitrification of human oocyte in medium supplemented with Latrunculin A
  Arms: Latrunculin A supplemented vitrification medium

SUMMARY:
Using cytoskeleton Stabilizer the Latrunculin A would improve the outcome of oocyte vitrification

ELIGIBILITY:
Inclusion Criteria:

* indication for oocyte cryopreservation

Exclusion Criteria:

-

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
survival after thawing | 6 days after thawing

SECONDARY OUTCOMES:
fertilization rate | 6 days of culture
Rates of blastocyst formation and quality | 6 days of culture
  Number of formed blastocyst and high-quality blastocysts per fertilized oocytes
embryo utilization rate | 6 days of culture
  Number of utilized embryos per fertilized oocytes
clinical pregnancy rate | three months
  Number of pregnant women with fetal pulsation per recruited cycles
ongoing pregnancy rate | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, IbnSina Hospital, Sohag